CLINICAL TRIAL: NCT01274689
Title: External Lid Loading for the Temporary Treatment of the Paresis of the M. Orbicularis Oculi: a Clinical Note
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Medical Park AG (Industry)
Other Study IDs: NCT100111
Record Dates: First submitted 2011-01-10; First posted 2011-01-11 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2008-06

CONDITIONS: Incomplete Closure of Lid; Parotis Tumor; m. Orbicularis Oculi Paresis
Keywords: lagophthalmos; parotis tumor; m. orbicularis oculi paresis
MeSH Terms: conditions — Lagophthalmos

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cohort: cohort of consecutively enrolled patients with lagophthalmos
  Interventions: Other: individually tailored lead weight

INTERVENTIONS:
Other: individually tailored lead weight — patients were treated with an individually tailored lead weight to train M. orbicularis oculi during day time

SUMMARY:
The note re-introduces the external lid loading with the help of a lead weight for the temporary treatment of lagophthalmos. Although simple and effective, the technique is rarely used.Instead of wearing a monoculus, the patient uses an individually tailored lead weight (0.8 mm thickness, 1.0 -2.0 g) sticked on the lid, it enables its closure. A spontaneous ptosis indicates a too heavy weight. With the M. levator palpebrae intact, lid lifting is possible. The effect is gravity dependent, so that the patient has to wear the monoculus at night. To minimize the risk of lead intoxication, the surface of the weight is varnished. In case of a persistent paresis of the M. orbicularis oculi an internal lid loading can follow. A total of 152 lagophthalmos cases have been treated since 1997.All patients could close the lid immediately. Almost half of the patients had to re-adjust the weight several times per day due to hooded eyelids. The compliance was high, and a partial or complete restoration of the function of the M. orbicularis oculi occurred in 60% of the cases. In some subjects, the restoration of the M. orbicularis oculi was faster than of the M. orbicularis orbis. The external lid loading for the temporary treatment of lagophthalmos is simple and effective. Compared to a monoculus, the vision is unimpaired and the aesthetic is more appropriate for most patients. The faster restoration of the M. orbicularis oculi hints at a potentially facilitatory effect of the weight.

ELIGIBILITY:
Inclusion Criteria:

* lagophthalmos due to surgery, central or peripheral paresis able to understand the purpose of the study

Exclusion Criteria:

* skin irritations and/or open wounds in the area of the applied lead weight

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with lagophthalmos due to surgery, central or peripheral paresis
Sampling Method: Non-Probability Sample
Enrollment: 152 (Estimated)
Dates: Start 1997-05; Primary Completion 2010-05 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
responder lid closure
  responder was created, whether the lid closure was a) not possible, b) partially possible, c) completely possible

SECONDARY OUTCOMES:
skin irritation
  was there a skin irritation after applicating the lead weight; yes or no

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Hesse, MD, Principal Investigator — Charite - University Medicine Berlin, Medical Park Berlin
Locations (1):
- Charité University Medicine Berlin, Medical Park Berlin, Berlin, State of Berlin, Germany

REFERENCES:
- [Background] Muller-Jensen K, Muller-Jensen G. [Surgical and conservative treatment of lagophthalmus (facial paralysis). II]. Ophthalmologe. 1993 Feb;90(1):27-30. German. PMID 8443444